CLINICAL TRIAL: NCT05270837
Title: A Phase 3 Multi-Center Study to Evaluate the Safety and Efficacy of Subcutaneous Injections of Pegvaliase in Adolescent Subjects (Ages 12-17) With Phenylketonuria Featuring an Open-Label Randomized Two-Arm (Active vs Diet-Only Control) Design
Brief Title: Study to Evaluate the Safety and Efficacy of Pegvaliase in Adolescents (Ages 12-17) With Phenylketonuria
Acronym: PEGASUS
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 165-306
Record Dates: First submitted 2022-02-01; First posted 2022-03-08 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Phenylketonuria (PKU)
Keywords: PKU; BioMarin; Phenylketonuria; BMN165; PAL; Subcutaneous Injections; Pegvaliase; adolescent PKU
MeSH Terms: conditions — Phenylketonurias | interventions — pegvaliase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pegvaliase (Experimental)
  Interventions: Drug: Pegvaliase
- Diet Only (Other): Participants will be managing their PKU with diet alone. Participants in the diet-only control arm will be required to maintain and adjust dietary and medical protein food intake through Week 72, initiating pegvaliase treatment beginning Week 73 and, from Weeks 73 through 215.
  Interventions: Other: Diet Only

INTERVENTIONS:
Drug: Pegvaliase — Pegvaliase 2.5mg/10mg/20mg/40mg/60mg self-administered from 1 time up to 7 times a week
  Other Names: PEG PAL; BMN 165
  Arms: Pegvaliase
Other: Diet Only — Diet Control
  Arms: Diet Only

SUMMARY:
This is a Phase 3 open-label randomized controlled study enrolling approximately 54 adolescents with PKU. The study is designed to assess the safety and efficacy of pegvaliase injections.

DETAILED DESCRIPTION:
This Phase 3 multicenter study is designed to evaluate the safety and efficacy of pegvaliase administered daily to adolescents (ages 12 to 17 years old (US), inclusive, and 12 to 15 years old (EU), inclusive 12-17) with phenylketonuria (PKU). Participants will be randomized in a 2:1 ratio to the active (pegvaliase) and control (diet-only) treatment arms, respectively, with 36 participants receiving pegvaliase and 18 participants managing their PKU with diet alone.

ELIGIBILITY:
Inclusion Criteria

* Is 12 to 17 years old (US), inclusive, or 12 to 15 years (EU), inclusive, at the start of the Screening/Run-in Period (Day -28).
* Diagnosis of PKU and failure to maintain recommended blood Phe levels on existing management (sapropterin dihydrochloride and Phe-restricted diet) demonstrated by 2 blood Phe concentration measurements > 600 μmol/L during the Screening/Run-in Period (7 to 10 days in between blood Phe assessments) and average blood Phe concentration > 600 μmol/L over the past 12 months (per available data).
* Willing and able to maintain and adjust dietary and medical protein food intake according to the study protocol under the supervision of a study dietician or adequately trained designee per investigator discretion during study participation.
* If on medication for ADHD, depression, or other psychiatric disorder, stable dose of medication for ≥ 8 weeks prior to enrollment and willing to maintain stable dose unless a change is medically indicated.
* An adult (≥ 18 years of age) has been identified who is willing and competent to observe the participant during study drug administration and for a minimum of 1 hour following administration.
* Participants must be capable of giving signed informed consent
* If sexually active, male or female participants must not plan to become pregnant (self or partner) and must use 2 acceptable methods of contraception while participating in the study beginning at Screening and for 4 weeks after discontinuing study drug.

Exclusion Criteria

* Previous treatment with pegvaliase.
* Use of any medication that is intended to treat PKU, including the use of large neutral amino acids, within 14 days prior to the administration of study drug on Day 1.
* Use or planned use of any injectable drugs containing polyethylene glycol (PEG; other than pegvaliase), including medroxyprogesterone injection, within 3 months prior to the start of Screening/Run-in and during study participation with the exception of COVID-19 vaccinations.
* A history of organ transplantation or on chronic immunosuppressive therapy.
* Use of any investigational product or investigational medical device within 30 days prior to Screening/Run-in or requirement for any investigational agent prior to completion of all scheduled study assessments.
* A positive test for HIV antibody, hepatitis B surface antigen, or hepatitis C antibody.
* Alanine aminotransferase (ALT) concentration > 2 × the upper limit of normal (ULN).
* Creatinine > 1.5 × ULN.
* Inability to identify and/or communicate to others that the participant is experiencing symptoms of potential anaphylaxis due to cognitive impairment or other reasons.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 55 (Estimated)
Dates: Start 2022-06-17 (Actual); Primary Completion 2025-01-14 (Actual); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Change in blood Phe concentration | Treatment naïve baseline following 72 weeks on study
Incidence of treatment-emergent adverse events as assessed by CTCAE v5.0 | Treatment naïve baseline following 72 weeks on study

SECONDARY OUTCOMES:
Change in total dietary protein intake | Treatment naïve baseline following 72 weeks on study

OTHER OUTCOMES:
Characterize area under plasma concentration time curve (AUC) of pegvaliase | Baseline to 215 weeks
Characterize maximum plasma concentration (Cmax) of pegvaliase | Baseline to 215 weeks
Characterize trough plasma concentration (Ctrough) of pegvaliase | Baseline to 215 weeks
Characterize time to reach maximum plasma concentration (Tmax) of pegvaliase | Baseline to 215 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Chair — BioMarin Pharmaceutical
Locations (16):
- United States (13):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Children's Hospital of Colorado, Aurora, Colorado
  - University of South Florida, Tampa, Florida
  - Ann and Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - IU Health University Hospital, Indianapolis, Indiana
  - University of Kentucky College of Medicine, Lexington, Kentucky
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - McGovern Medical School, University of Texas Health Science Center at Houston (UTHealth), Houston, Texas
  - University of Utah Medical Center, Salt Lake City, Utah
  - University of Virginia School of Medicine, Charlottesville, Virginia
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Germany (3):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Universitat Mainz, Mainz